CLINICAL TRIAL: NCT00657358
Title: The Effect of Intravenous Lidocaine on Normal Sensation and Pain in Healthy Volunteers (Carl Koller Grant) (The Effect of Intravenous Lidocaine on Allodynia)
Brief Title: The Effect of Intravenous Lidocaine on Normal Sensation and Pain in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: American Society of Regional Anesthesia (Other)
Responsible Party: Principal Investigator, Michael Froelich, Michael A. Froelich, M.D., University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F061204013
Record Dates: First submitted 2008-04-09; First posted 2008-04-14 (Estimated); Results first posted 2014-01-13 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-04

CONDITIONS: Pain
Keywords: lidocaine; allodynia; chronic regional pain syndrome; pain
MeSH Terms: conditions — Pain; Hyperalgesia; Complex Regional Pain Syndromes | interventions — Lidocaine; Anesthesia, Local

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lidocaine (Experimental): Lidocaine 2% (2mg/ml) was administered via a computer assisted infusion to achieve a target plasma concentration of 2 mcg/ml; infused within 20 minutes.
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — Lidocaine 2% (2mg/ml) was administered via a computer assisted infusion to achieve a target plasma concentration of 2 mcg/ml; infused within 20 minutes.
  Other Names: Local Anesthesia

SUMMARY:
The purpose of this study is to study if lidocaine, given intravenously, reduces pain.

DETAILED DESCRIPTION:
Clinicians use lidocaine intravenously in a fashion that suggests that it might have analgesic effects. Therefore, we test the hypothesis that lidocaine reduces pain intensity in response to experimental pain.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Adult Volunteers, age >19 years

Exclusion Criteria:

* History of Substance Abuse
* Coronary Artery Disease (CAD): unstable
* Congestive Heart Failure (CHF): unstable
* Heart Arrhythmia: symptomatic
* Chronic Obstructive Pulmonary Disease (COPD)
* Lidocaine Allergy
* Diagnostic and Statistical Manual of Mental Disorders (Rev IV): Axis I: Common Axis I disorders include depression, anxiety disorders,bipolar disorder, ADHD, and schizophrenia. Axis II: borderline personality disorder, schizotypal personality disorder, antisocial personality disorder, and mild mental retardation.
* Presence of Contraindications for MRI
* Presence of electronically, magnetically, and mechanically activated implants
* Electronically, magnetically, and mechanically activated implants
* Ferromagnetic or electronically operated active devices like automatic cardioverter defibrillators
* Cardiac pacemakers
* Metallic splinters in the eye
* Ferromagnetic haemostatic clips in the central nervous system (CNS)
* Claustrophobia
* Pregnancy

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-04; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Froelich, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Lidocaine: Healthy Volunteers receiving Lidocaine
Period: Overall Study
Arm/Group | Lidocaine
Started | 22
Completed | 16
Not Completed | 6
Not completed — Lack of Efficacy | 6

BASELINE CHARACTERISTICS:
Arm/Group | Lidocaine
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Ischemic Pain
Description: The right arm was exsanguinated by elevating it above heart level for 30 seconds, after which the arm was occluded with a standard blood pressure cuff positioned proximal to the elbow inflated to twice the participant's mean arterial pressure. Participants then performed 20 handgrip exercises of 2-second duration at 4-second intervals at 50% of their maximum grip strength. Pain was rated on a scale from 0 - 10 with 0 being no pain to 10 being the worst pain imaginable.
Time Frame: baseline, during 20 minute lidocaine infusion, and 30 minutes after discontinuation of lidocaine infusion
Population: health volunteers
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Lidocaine Administration: Lidocaine 2% (2mg/ml) was administered via a computer assisted infusion to achieve a target plasma concentration of 2 mcg/ml; infused within 20 minutes.
Arm/Group | Lidocaine Administration
Number analyzed (Participants) | 16
units on a scale
  Baseline (prior to administration) | 4.31 (.48)
  During 20 Infusion | 3.49 (.48)
  30 After Infusion completed | 3.44 (.48)
Statistical Analysis 1: Comparison: Lidocaine Administration; Test type: Superiority or Other; p < 0.001, Regression, Linear; DF=2 DFDEN=371.8, F-ratio=10.66; R^2 (adj) = 0.477

2. Primary Outcome: Electrical Pain
Description: Peripheral nerve stimulation electrodes were attached to the base and the tip of the third digit and connected to a constant current stimulator (DS7A, Digitimer Ltd, Hertfordshire, England). Ascending electrical stimuli of 2000 mu duration, ranging from 0.5 to 35 mA (ampere) was administered one per second in 0.5 mA increments. Participants were instructed to indicate when they first felt the slightest sense of pain (electrical pain threshold, EPTh) and when they were unable to tolerate a further increase (electrical pain tolerance, EPTo). For each measure, the average of three trials was computed for use in subsequent analyses. Each of the three electrical pain stimuli were presented three times and balanced in order using a Graeco-Latin square design. The pain scale is between 0 and 10, with 0 being no pain and 10 being the worst pain imaginable
Time Frame: Baseline, during 20 minutes lidocaine infusion, and 30 minutes after completion of lidocaine infusion
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Lidocaine Administration: Lidocaine 2% (2mg/ml) was administered via a computer assisted infusion to achieve a target plasma concentration of 2 mcg/ml; infused within 20 minutes.infused within 20 minutes.
Arm/Group | Lidocaine Administration
Number analyzed (Participants) | 16
units on a scale
  Baseline - at time of lidocaine administration | 2.40 (0.34)
  During 20 minute lidocaine Infusion | 2.04 (.34)
  30 minutes after compleition of lidocaine infusion | 2.52 (.34)

3. Primary Outcome: Heat Pain
Description: The thermal procedure involved a baseline assessment of heat pain threshold and tolerance. Contact heat stimuli were delivered using a computer-controlled Medoc Thermal Sensory Analyzer (TSA-II; Ramat Yishai, Israel), which is a peltier elementbased stimulator. Temperature levels were monitored by a thermistor and returned to a preset baseline of 32°C by active cooling at a rate of 10°C/s. The 3 × 3 cm contact probe was applied to the right forearm. The pain scale is between 0 and 10 with 1 being no pain and 10 being the worst pain imaginable
Time Frame: baseline, during 20 minute lidocaine infusion, and 30 minutes after completion of lidocaine infusion
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Lidocaine Administration
Number analyzed (Participants) | 16
units on a scale
  Baseline - at start of lidocaine infusion | 3.01 (0.42)
  During 20 minute lidocaine infusion | 2.83 (.42)
  30 minutes after completion of lidocaine infusion | 2.82 (.42)

4. Primary Outcome: Cold Pain
Description: The participant's foot was immersed up to the ankle into a container filled with ice water of 3°C. Participants were instructed to maintain their foot in the container until the cold pain became intolerable (cold pain tolerance). The length of time was recorded in seconds. This procedure was repeated once with a gap of at least fifteen minutes in-between repeated tests. The range was 0 seconds to 120 seconds
Time Frame: baseline, during 20 minute infusion, and 30 minutes after lidocaine infusion
Measure: Mean (Standard Error); unit: time in seconds to withdrawal
Arm/Group | Lidocaine Administration
Number analyzed (Participants) | 16
time in seconds to withdrawal
  Baseline - at start of infusion | 42 (10.9)
  During 20 minute lidocaine infusion | 50.6 (10.9)
  30 minutes after completion of lidocaine infusion | 51.2 (11.0)

5. Primary Outcome: Tactile Sensation
Description: Pin prick sensory thresholds (PPT) were obtained by touching the skin in-between the first and second metacarpal bone with a 23-gauge needles which moved freely out of a 10 mL plastic syringe barrel. The pin prick sensation was modified by adding small weights to the 23-gauge needles (from 0.2 to 5.2 mg). A syringe barrel of tuberculin (TB) needles that were cut to different lengths to add the desired weight to the 23-gauge needle. The PPT was determined using the weighted 23-gauge needle in ascending order, according to the method of limits. This assessment was to evaluate whether participants were able to feel the touch of the needle. The participant's arm was placed on a tray table. A linen sheet was suspended in-between two IV poles in such a fashion that the subject's view of his/her hand was blocked. Normal values are between 0.21mg and 5mg.
Time Frame: baseline, during 20 minute infusion, and 30 minutes after completion of infusion
Measure: Mean (Standard Error); unit: weight in mg
Arm/Group | Lidocaine Administration
Number analyzed (Participants) | 16
weight in mg
  Baseline - at start of lidocaine administration | .28 (.02)
  During 20 minute Infusion | .27 (.02)
  30 Minutes after completion of infusion | .27 (.02)

ADVERSE EVENTS:
Arm/Group | Lidocaine
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Restriction type: embargo of more than 60 days